CLINICAL TRIAL: NCT07022886
Title: INCIDENCE, PREVALENCE AND OVERALL RISK OF ESOPHAGEAL CANCER IN ACHALASIA: A PROPENSITY-MATCHED POPULATION-BASED STUDY FROM A LARGE MULTICENTER DATABASE
Acronym: RECAP
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Collaborators: TriNetX, LLC (Unknown); Vita-Salute San Raffaele University (Unknown)
Responsible Party: Principal Investigator, Alberto Barchi, Medical Doctor, IRCCS San Raffaele
Other Study IDs: RECAP
Record Dates: First submitted 2025-06-08; First posted 2025-06-15 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Achalasia Cardia; Esophageal Cancer (EsC)
Keywords: achalasia; esophageal cancer
MeSH Terms: conditions — Esophageal Achalasia; Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Achalasia primary cohort: Achalasia cohort (both naive or treated)
- Control subjects: Healthy controls, with the exclusion of achalasia
- Achalasia without Barrett Esophagus: Sensitivity analysis of achalasia both treated or untreated without Barrett esophagus
- Treated achalasia: achalasia undergone to various treatments
  Interventions: Procedure: achalasia treatments
- Untreated achalasia: Achalasia without previous treatment
- LHM: Heller-Dor myotomy
  Interventions: Procedure: achalasia treatments
- POEM: Peroral endoscopic myotomy
  Interventions: Procedure: achalasia treatments

INTERVENTIONS:
Procedure: achalasia treatments — esophageal achalasia treatments
  Other Names: POEM; LHM
  Groups: LHM; POEM; Treated achalasia

SUMMARY:
Esophageal Achalasia has been investigated as a potential risk factor for esophageal cancer (EC). Longstanding disease, repeated treatment, age and male sex seem the most relevant risk factors, but no clear effect size estimation from large sample cohorts has been provided so far. The aim of the investigators is to estimate EC risk in large sample-size population, and to provide sub-analyses per cancer type and treatment impact on EC risk.

DETAILED DESCRIPTION:
Achalasia is a chronic idiopathic condition characterized by the absence of esophageal peristalsis and reduced relaxation of the lower esophageal sphincter, causing progressive dysphagia and weight loss. Achalasia has been investigated as a potential risk factor for esophageal cancer (EC); squamous cancer due to chronic inflammation related to stasis due to poor esophageal emptying and adenocarcinoma due to uncontrolled gastroesophageal reflux after treatment. Longstanding disease, repeated treatment, age and male sex have been addressed as the most relevant risk factors, but no clear effect size estimation from large sample cohorts has been provided so far.

The authors conducted a retrospective cohort study, accessing the global federated health research network "TriNetX", that provides access to electronic medical records from approximately a hundred million patients across large healthcare organizations (HCOs). The analysis will be performed on achalasia patients, based on the ICD-10 code (K22.0), from January 1st 2000 until May 31st 2025. The incidence rate (cases/1000 persons-year) and cumulative prevalence of EC in an achalasia cohort in a span of 25 years will be firstly assessed. Then the absolute and time-to-event risk of EC, by comparing the achalasia cohort with control cohort, after propensity score nearest neighbor greedy matching, for relevant covariates. Kaplan-Meyer (KM) analysis with censoring, Hazard Ratios (HRs) and Risk Ratio (RR) and Risk Difference (RD) estimation for EC risk will be calculated. Log Rank test will be used to compare KM curves. Further sub-group analysis will be implemented between two population of achalasia patients, treated (with endoscopic/surgical myotomy or pneumatic dilation) and treatment-naïve. Further in-depth analyses between histologic type of EC, esophageal localization and comparing different achalasia treatment (myotomy vs pneumatic dilation) will be performed, in order to categorize the risk of EC, if more linked to treatment and therefore to the development of reflux, Barrett esophagus eventually leading to adenocarcinoma, or towards squamous cell cancer driven by chronic stasis and degeneration of the squamous esophageal epithelium

ELIGIBILITY:
Inclusion Criteria:

* Esophageal achalasia diagnosed according to guidelines (ICD-10-K22.0)

Exclusion Criteria:

* Primary esophaeal and pharyngeal motility disorders (ICD-10-J39.2)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Achalasia diagnosis according to guidelines as stated in Electronic Health Records (EHR) data.
Sampling Method: Non-Probability Sample
Enrollment: 47000 (Actual)
Dates: Start 2025-06-03 (Actual); Primary Completion 2025-06-03 (Actual); Study Completion 2025-09-07 (Estimated)

PRIMARY OUTCOMES:
Hazard Ratio | from Jan 1st 2000 to June 3rd 2025
  Hazard Ratio (HR) with Kaplan Meyer (KM) analysis of EC occurrence in achalasia vs control subjects
Incidence proportion, prevalence and incidence rate | Jan 1st 2000- June 3rd 2025
  Incidence proportion (%), prevalence (%) and incidence rate (100,000 persons-year) of EC (and different histological subtypes)

SECONDARY OUTCOMES:
Risk Ratio | Jan 1st 2000-Jun 3rd 2025
  Risk Ratio of EC (and different histologic subtypes) occurrence in achalasia cohort compared to controls, in treated vs untreated achalasia, LHM vs POEM group
Risk Difference | Jan 1st 2000-June 3rd 2025
  Risk Difference of EC (and different histological subtypes) occurrence in achalasia cohort compared to controls, in treated vs untreated achalasia, LHM vs POEM group
Hazard Ratio (HR) with Kaplan Meyer (KM) analysis of EC occurrence | Jan 1st 2000- June 3rd 2025
  Hazard Ratio (HR) with Kaplan Meyer (KM) analysis of EC occurrence (according to different subtypes) in achalasia vs control subjects and in treated vs untreated achalasia, and in LHM vs POEM

CONTACTS AND LOCATIONS:
Overall Officials: Albert Jan Bredenoord, MD, PhD, Prof, Study Director — Department of Gastroenterology, Amsterdam UMC Location AMC, Amsterdam, The Netherlands
Locations (1):
- IRCCS San Raffaele Hospital, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
No IPD used in this study

REFERENCES:
- [Background] Ponds FA, Moonen A, Smout AJPM, Rohof WOA, Tack J, van Gool S, Bisschops R, Bredenoord AJ, Boeckxstaens GE. Screening for dysplasia with Lugol chromoendoscopy in longstanding idiopathic achalasia. Am J Gastroenterol. 2018 Jun;113(6):855-862. doi: 10.1038/s41395-018-0064-1. PMID 29748564
- [Background] Tustumi F, Bernardo WM, da Rocha JRM, Szachnowicz S, Seguro FC, Bianchi ET, Sallum RAA, Cecconello I. Esophageal achalasia: a risk factor for carcinoma. A systematic review and meta-analysis. Dis Esophagus. 2017 Oct 1;30(10):1-8. doi: 10.1093/dote/dox072. PMID 28859394
- [Background] Gillies CL, Farrukh A, Abrams KR, Mayberry JF. Risk of esophageal cancer in achalasia cardia: A meta-analysis. JGH Open. 2019 Feb 8;3(3):196-200. doi: 10.1002/jgh3.12132. eCollection 2019 Jun. PMID 31276035
- See also: TriNetX platform link — https://live.trinetx.com/